CLINICAL TRIAL: NCT05130957
Title: The Effect of Massage Applied With Clove Oil on Perceived Labor Pain
Brief Title: The Effect of Clove Oil on Labor Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Nükhet Kaçar, Principal Investigator, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AnkaraCHBilkent-MH-NK-01
Record Dates: First submitted 2021-11-12; First posted 2021-11-23 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Labor Pain
Keywords: labor pain; midwifery; pregnant women; massage
MeSH Terms: conditions — Labor Pain | interventions — Clove Oil

STUDY DESIGN:
Intervention Model Description: There are two groups as experimental and control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): The pregnant women in the experimental group are given a massage with clove oil.
  Interventions: Other: Massage Application with clove oil
- Control Group (Other): The pregnant women in the control group are given a massage without any oil as standard midwifery care
  Interventions: Other: Massage Application without any oil

INTERVENTIONS:
Other: Massage Application with clove oil — The experimental group is given a massage with clove oil,
  Arms: Experimental Group
Other: Massage Application without any oil — The control group is given a massage without any oil as a standard midwifery care.
  Arms: Control Group

SUMMARY:
The study has two groups. one of them is experimental group that is given massage with clove oil. The other one is control group that is given standard midwifery care. Each group consists of 30 women. We will evaluate their labor pain scores by using Visual Analogue Scale before and after massage application.

DETAILED DESCRIPTION:
Labor is a painful process. That's why there are lots of nonpharmacological methods to reduce labor pain. Especially most clinical guide suggests giving massage to pregnant who has labor pain. In the literature, there are a lot of study examining effectiveness of massage techniques. However there is no study about massage application with clove oil on labor pain. The investigators would like to give a massage with clove oil to pregnants to reduce their labor pain. Hereby the investigators will evaluate effectiveness of clove oil.

ELIGIBILITY:
Inclusion Criteria:

* All of volunteer and pregnant women is 18-35 years old.

Exclusion Criteria:

* The pregnant women has any obstetrical complications.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Because we study with pregnant women
Enrollment: 60 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | during labor process, until the labor process is done.
  The scale has 0-10 points. As the point increases the pain score increases

CONTACTS AND LOCATIONS:
Overall Officials: Nükhet Kaçar, MSc., Principal Investigator — Ankara City Hospital- Maternity Hospital
Locations (1):
- Ankara City Hospital- Maternity Hospital, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No